CLINICAL TRIAL: NCT05738525
Title: Comparative Study of Automated Peritoneal Dialysis With Remote Patient Management And Continuous Ambulatory Peritoneal Dialysis on the Prognosis and QOL in Peritoneal Dialysis Patients
Brief Title: Comparative Study of Prognosis and QOL Between APD-RPM and CAPD
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Professor, Chief physician, Academician of Chinese Academy of Engineering, Chinese PLA General Hospital
Other Study IDs: S2022-775-01
Record Dates: First submitted 2023-02-09; First posted 2023-02-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: End-stage Renal Disease
Keywords: APD-RPM; CAPD; Prognosis; QOL; Comparative Study
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Automated peritoneal dialysis with remote patient management (APD-RPM): APD mode is recommended but not limited to continuous circulating peritoneal dialysis (CCPD). Dialysis dose ranges from 5 to 10 liters per day and glucose concentration starts from low concentration (1.5%).
  Interventions: Device: APD-RPM
- Continuous ambulatory peritoneal dialysis (CAPD): (1) Dialysis dose ranges from 5 to 10 liters per day at the run-in period. For those with regular peritoneal dialysis, the original dose can be used according to the volume status and solute clearance effect in the past 3 months; (2) Exchange time and abdominal retention time is generally 2-5 times and 1 time at daytime and night, separately; (3) Glucose concentration includes 1.5%, 2.5% or 4.25%; (4) The treatments can be adjusted according to the change of residual renal function, peritoneal transport characteristics, volume status, solute clearance, clinical status and peritonitis.

INTERVENTIONS:
Device: APD-RPM — APD mode is recommended but not limited to continuous circulating peritoneal dialysis (CCPD); (2) Dialysis dose ranges from 5 to 10 liters per day and depends on previous APD prescription and dialysis adequacy; (3) Glucose concentration starts from low concentration (1.5%) and depends on previous dialysis prescription.
  Remote monitoring includes dynamic changes of the overall treatment situation, warning or any abnormal notes, and drainage, retention and duration of APD per day.
  Groups: Automated peritoneal dialysis with remote patient management (APD-RPM)

SUMMARY:
This is an observational, multicenter, parallel control study, planning to enroll 750 eligible patients to receive automated peritoneal dialysis with remote patient management (APD-RPM) and continuous ambulatory peritoneal dialysis (CAPD). Patients will attend follow-up every 12 ± 1 weeks for a total of 156 weeks. This study aims to compare the effects of APD-RPM and CAPD treatment on the prognosis and quality of life.

DETAILED DESCRIPTION:
This is an observational study based on the real-word diagnosis and treatments. Target subject population include end-stage renal disease patients (aged 18-75 years) with peritoneal dialysis 3 months and longer. Standard peritoneal balance test of eligible patients should be rapid peritoneal solute transfer rate (4-hour D/P creatinine value > 0.65). Patients will be divided into two groups to receive standard APD-RPM or CAPD with a ratio of 1:2.

Peritoneal dialysis in APD-RPM group (n=250): (1) APD mode is recommended but not limited to continuous circulating peritoneal dialysis (CCPD); (2) Dialysis dose ranges from 5 to 10 liters per day and depends on previous APD prescription and dialysis adequacy; (3) Glucose concentration starts from low concentration (1.5%) and depends on previous dialysis prescription.

Peritoneal dialysis in CAPD group (n=500): (1) Dialysis dose ranges from 5 to 10 liters per day at the run-in period. For those with regular peritoneal dialysis, the original dose can be used according to the volume status and solute clearance effect in the past 3 months; (2) Exchange time and abdominal retention time is generally 2-5 times and 1 time at daytime and night, separately; (3) Glucose concentration includes 1.5%, 2.5% or 4.25%; (4) The treatments can be adjusted according to the change of residual renal function, peritoneal transport characteristics, volume status, solute clearance, clinical status and peritonitis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years to 75 years
* Confirmed diagnosis of end-stage renal disease
* Standard peritoneal balance test shows rapid peritoneal solute transfer rate, defined as 4 hours D/P creatinine value greater than 0.65
* Be able to comply with the standard peritoneal dialysis treatment at home
* Peritoneal dialysis time 3 months and longer
* Fully understand the study and have signed the informed consent

Exclusion Criteria:

* Prepare for kidney transplantation within 3 years
* Need combined treatment of hemodialysis
* Be allergic to components of peritoneal dialysis fluid
* Complicated with severe cardio-cerebrovascular diseases such as congestive heart failure, grade III and above of NYHA classification, acute myocardial infarction within 3 months, malignant arrhythmia requiring treatment, dilated cardiomyopathy, acute cerebral infarction or acute cerebral hemorrhage within 3 months, etc.
* Complicated with serious liver diseases, such as cirrhosis or acute liver injury [Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) 2 times greater the the normal]
* Active or treated residual malignant tumors, HIV infection
* Pregnant or lactating women at childbearing age who disagree to use effective contraceptives during the trial
* History of alcohol or drug (illegal drugs) abuse
* Unable to continue CAPD due to ultrafiltration failure
* Mental retardation or mental illness
* Patients who use icodextrin dialysate
* Participation in other clinical trials in the past 3 months
* Peritonitis in the past 3 months
* Other situations decided by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 750 patients with end-stage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause deaths/technical failure | 156 weeks from baseline
  The time from baseline to all-cause death or technical failure
Quality of life (QOL) | 156 weeks from baseline
  Change of quality of life (QOL) score from the baseline
Returning to society | 156 weeks from baseline
  Change of assessment of returning to society from the baseline

SECONDARY OUTCOMES:
Cardio-cerebrovascular events | Up to 156 weeks
  Incidence of cardio-cerebrovascular events, including sudden cardiac death, serious arrhythmia, coronary heart disease requiring interventional treatment, congestive heart failure with grade III and above of New York Heart Association (NYHA) classification, acute cerebral infarction, and acute cerebral hemorrhage
Ultrafiltration rate | Up to 156 weeks
  Change of ultrafiltration rate from baseline
Capacity overload | Up to 156 weeks
  Degree, proportion and frequency of capacity overload
Hypertension and antihypertension drugs | Up to 156 weeks
  Proportion of well-controlled hypertension. Quantity of antihypertension drugs
Peritonitis | 156 weeks from baseline
  Proportion of peritonitis. Time to first peritonitis from enrollment
Glomerular Filtration Rate | Up to 156 weeks
  Change of slope of renal function Glomerular Filtration Rate (GFR)
Nutritional status | 24, 48, 72, 96 120, 144, 156 week
  Change of subjective global assessment (SGA) score from baseline
Adequacy of dialysis | Up to 156 weeks
  Proportion of adequacy of dialysis
Prescription adjustment, outpatient follow-up and unplanned outpatient visits | Up to 156 weeks
  Times of prescription adjustment, outpatient follow-up and unplanned outpatient visits
Hospitalization | Up to 156 weeks
  Proportion of hospitalization and unplanned hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Xiangmei Chen, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China